CLINICAL TRIAL: NCT00447213
Title: A Crossover Study to Evaluate the Efficacy and Safety of Preprandial Human Insulin Inhalation Powder (HIIP) Compared to Preprandial Injectable Insulin in Patients With Type 1 Diabetes Mellitus
Brief Title: A Study for Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Alkermes, Inc. (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10299; H7U-JE-IDBB
Record Dates: First submitted 2007-03-12; First posted 2007-03-14 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Insulin glargine; Drug: Human Insulin Inhalation Powder; Drug: Injectable Insulin
- 2 (Experimental)
  Interventions: Drug: Insulin glargine; Drug: Human Insulin Inhalation Powder; Drug: Injectable Insulin

INTERVENTIONS:
Drug: Insulin glargine — Patient specific, injected, daily, 24 weeks
Drug: Human Insulin Inhalation Powder — patient specific dose, inhaled, before meals,12 weeks
  Other Names: LY041001
Drug: Injectable Insulin — Patient specific dose,injected, before meals, 12 weeks

SUMMARY:
The purpose of the study is to compare the human insulin inhalation powder plus insulin glargine with injected insulin (regular human insulin or insulin lispro) plus insulin glargine on lowering the blood sugar level.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus for at least 24 months
* Injecting insulin (insulin lispro, aspart or regular insulin, insulin lispro/aspart mixtures, or regular human insulin mixtures) in the last 24 months
* HbA1c equal or less than 11 %
* Nonsmokers, had not smoked for at least 6 months and agree not to smoke (cigars, cigarettes or pipes) or use smokeless tobacco for the duration of the study
* Satisfactory lung function results to meet the requirement of the study

Exclusion Criteria:

* Previously received any form of inhaled insulin
* Require a daily total insulin dosage greater than 100 U
* Have a current or past history of asthma, chronic obstructive pulmonary disease or other clinically relevant lung disease
* History or presence of liver disease
* History or presence of kidney disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline | 12 and 24 weeks

SECONDARY OUTCOMES:
Proportion of patients who achieve an HbA1c < 7% and <= 6.5% | 12 and 24 weeks
Insulin (regular human insulin, insulin lispro, human insulin inhalation powder or insulin glargine)doses | at each visit
8-point self monitoring blood glucose profiles | 12 and 24 weeks
Two hour glucose excursions for the morning, midday, and evening meals | 12 and 24 weeks
Inhaler reliability | throughout the study
Patient-reported treatment satisfaction and insulin delivery satisfaction | 12 and 24 weeks
Preference for the study therapies | week 24

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-277-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- Japan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- Taiwan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changhua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taoyuan District

REFERENCES:
- [Result] Hitoshi Ishii, Satoru Tsujii, Masami Tanaka, Miyuki Furuya, Tadao Iburi, Rei Ueda, Sakura Okuyama, Risa P. Hayes, Masato Okamura, Kazuya Iwamoto, Eisei Oda. Development of IDSQ-J and assessment of reproducibility adequacy. Tonyobyo. 2009;52(3):209-221.
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com